CLINICAL TRIAL: NCT01421901
Title: Antibiotics vs.Surgery in Acute Appendicitis;an Intention to Treat Prospective Randomised Study. The ASAA-study
Brief Title: Antibiotics Versus Surgery in Acute Appendicitis
Acronym: ASAA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Responsible Party: Principal Investigator, Michele Pisano, Medical Doctor, A.O. Ospedale Papa Giovanni XXIII
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EUDRA CT Number 2011-002977-44
Record Dates: First submitted 2011-08-04; First posted 2011-08-23 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Acute Appendicitis Without Peritonitis
Keywords: Acute appendicitis; Surgery; Antibiotics; comparison surgery and antibiotics; resolutions of symptoms
MeSH Terms: conditions — Appendicitis | interventions — Ertapenem; Appendectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ertapenem (Experimental)
  Interventions: Drug: Ertapenem
- appendectomy (Active Comparator): Appendectomy is compared to Ertapenem
  Interventions: Procedure: appendectomy

INTERVENTIONS:
Drug: Ertapenem — Ertapenem i.v,m 1g, once a day, 3 days
  Arms: Ertapenem
Procedure: appendectomy
  Arms: appendectomy

SUMMARY:
The acute appendicitis (AA) is a very common disease with a life time risk 7-8% and the highest incidence in the second decades . The aetiology of AA is still poor understood: the commonest hypothesis refers to appendix obstruction followed by impairment of wall appendix barrier and thus wall perforation and/or abscess formation1. However some studies suggest that no-complicate and complicate appendicitis are different entities allowing a different treatment. The study aims to test the no inferiority in terms of efficacy of antibiotic treatment compared to surgery in a population with high probability to suffer of 1st episode of AA.The study aims to test the no inferiority in terms of efficacy of antibiotic treatment compared to surgery in a population with high probability to suffer of 1st episode of AA.

ELIGIBILITY:
Inclusion Criteria:

* patients between 18 and 65 years old
* first episode of suspected AA diagnosed by Andersson's score or combination with abdominal ultrasound

Exclusion Criteria:

* patients with any potential immunodeficiency status
* assumption of antibiotics for different infectious disease or surgery in the last 30 days
* allergy to antibiotics established in the study protocol
* no acceptance of study protocol
* pregnancy or delivery in the last 6 months
* ASA IV or V, no Italian or English fluently speakers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2011-08; Primary Completion 2014-12 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
the rate of patients free of symptoms into 2 weeks (from operation in the surgery group or from the third Ertapenem administration in the antibiotics group) with no pain, no fever, WBC ≤ 10000, CRP ≤ 1 | 2 weeks

SECONDARY OUTCOMES:
Secondary outcomes will be considered major complications occurring after 2 weeks and into 1 year. Phone consultation will be performed at 1 year | 2 weeks- One year
  1. Surgery:
     Rate of reintervention due to bowel occlusion (idro fluid level at Abdomen xRay and/no resolution by Gasytograffin) or intraperitoneal abscess; incisional hernia or wound dehiscence.
  2. Antibiotic:
  Rate of Diagnosis of new AA. We will register also the rate of intervention for bowel occlusion longer than 48 hours (no passage of flatus, vomit or combination) or intraperitoneal abscess.
  Further secondary outcome are Wound infection, negative appendectomy. Hospital stay and work absence.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Ansaloni, Study Director — Papa Giovanni XXIII Hospital Bergamo; Michele Pisano, Principal Investigator — Papa Giovanni XXIII Hospital Bergamo
Locations (1):
- 1St General Surgery Unit Papa Giovanni XXIII Hospital Bergamo, Bergamo, Italy